CLINICAL TRIAL: NCT02480257
Title: University of California San Francisco (UCSF) TARA Study: Training for Awareness, Resilience and Action
Brief Title: UCSF TARA Study: Training for Awareness, Resilience and Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Edgewood Center for Children and Families (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-12380
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Depression; Anxiety
Keywords: intervention; emotion regulation; fMRI; mindfulness; yoga-based movement
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TARA Intervention group (Experimental): TARA is comprised of 12 weekly classes delivered in a group format by two trained facilitators with approximately 8-15 participants. The 90 minute sessions are designed to promote skills for autonomic regulation, attention modulation, emotion regulation and cognitive control.
  Interventions: Behavioral: TARA

INTERVENTIONS:
Behavioral: TARA — The intervention consists of four 3-week modules: 1. Autonomic regulation: Learning and practicing the ability to create a calm and safe inner state through breathing exercises and movement/physical activity. 2. Interoceptive awareness: Attention training, targeting external stimuli then sensory stimuli using short body scan exercises and guided meditations. 3.Emotion regulation: Recognizing, labeling, externalizing, and befriending emotions. 4. Metacognition, core-values, and committed action: Understanding social triggers to negative emotions and experiential avoidance strategies and their impact on obtaining desired life-goals. Home practice of TARA skills is encouraged, with breathing instructions and short, guided meditations provided via audio tracks.

SUMMARY:
The investigators aim to refine and pilot test an innovative group treatment model for adolescent depression and anxiety, Training for Awareness, Resilience and Action (TARA) in a sample of 14-18 year olds with depressive or anxious symptoms.

DETAILED DESCRIPTION:
The investigators aim to refine and pilot test an innovative group treatment model for adolescent depression and anxiety, Training for Awareness, Resilience and Action (TARA). TARA is based on our current understanding of the neuroscience of adolescent depression and anxiety. It employs specific approaches drawn from mindfulness practices and yoga to promote physiological regulation and attention modulation, emotion regulation, and cognitive control. The investigators will perform three initial (non-randomized) beta tests with 6-12 participants each to refine our intervention manual. The investigators will enroll up to 30 participants total, aged 14-18 with depression and/or anxiety symptoms, to receive the TARA intervention. The investigators hypothesize that TARA will be feasible in terms of recruitment, retention, adherence, and participant receptivity to the intervention as gauged through feedback surveys and a focus group. The primary outcomes are depression symptoms assessed with the Reynolds Adolescent Depression Scale (RADS-2) and anxiety symptoms assessed with the Multidimensional Anxiety Scale for Children (MASC). Secondary outcomes include self-reported emotion regulation and attention/awareness. The investigators hypothesize that participants will show improvements in these measures. In a small subset of participants, the investigators will also test the feasibility of using functional MRI (fMRI) before and after the intervention to measure the underlying neurobiological effects of TARA. The aim is to develop a protocol for possible future use in a larger study to examine effects of the intervention on patterns of amygdala activation linked with adolescent depression.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old, and not yet graduated from high school.
* Post-pubertal (Tanner Stage , stage 3+).
* CDRS-R score≥35 or MASC score≥56.
* Currently under the care of a physician or mental health provider for depression and/or anxiety.

Exclusion Criteria:

* Current comorbidity of psychosis, severe anorexia nervosa, PTSD, severe self-mutilation, severe suicidal ideation or attempt in past 3 mos.
* Comorbidity (lifetime) of bipolar disorder, low-functioning autism spectrum disorder, intellectual disability (estimated intelligence quotient < 80).
* A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the group intervention.
* Non English speaker.
* Current mindfulness training (e.g. Mindfulness Based Stress Reduction or Mindfulness Based Cognitive Therapy or Dialectical Behavior Therapy) and/or practice with a typically sitting meditation or yoga of 20 or more minutes two or more times per week for the past two months.
* Unable to attend study assessments and classes in San Francisco as scheduled.
* Special exclusion criteria will be applied for fMRI participation for safety reasons (pregnancy, claustrophobia, metallic implants); left-handedness; and for task performance (colorblindness or less than 20/40 correctable vision); not willing to abstain from alcohol and/or drugs for 2 weeks prior to the MRI . These participants can be included in the study but will be excluded from participation in fMRI.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reynolds Adolescent Depression Scale (RADS-2) | Change from 0 to 3 months
  Self report, 30-item measure of 4 dimensions of depression: Dysphoric Mood, Anhedonia/Negative Affect, Negative Self-Evaluation, and Somatic Complaints
Multidimensional Anxiety Scale for Children (MASC) | Change from 0 to 3 months
  Self report measure of anxiety,with 39 items distributed across four major factors, three of which can be parsed into two subfactors each. Main and subfactors include (1) physical symptoms (tense/restless and somatic/autonomic), (2) social anxiety (humiliation/rejection and public performance fears), (3) harm avoidance (perfectionism and anxious coping), and (4) separation anxiety.

SECONDARY OUTCOMES:
Children's Depression Rating Scale, Revised (CDRS-R) | 0, 3, and 6mos
  Standardized rating scale depression based on semi-structured interview. Seventeen symptom areas are assessed during the interview with a 5 or 7 point rating scale for each of the 17 domains. Each item is rated on a scale of 1 to 7, with 1 being least severe (no difficulties) to 7 indicating severe clinical difficulties. Domains assessed align with Diagnostic and Statistical Manual-IV (DSM-IV) criteria for childhood depression.
Insomnia Severity Index (ISI) | 0, 3, and 6 mos
  Self-report, 7-item assessment scale for sleeping problems.
Affective Reactivity Index (ARI) | 0, 3, and 6 mos
  Self-report, 6-item measure of irritability in children and teenagers.
The Avoidance and Fusion Questionnaire for Youth (AFQ-Y8) | 0, 3, and 6 mos
  8-item self-report measure of psychological inflexibility fostered by: (1) Cognitive fusion (2) Experiential avoidance (3) Inaction or behavioral ineffectiveness in the presence of unwanted internal experiences.
Child and Adolescent Mindfulness Measure (CAMM) | 0, 3, and 6 mos
  10-item self-report measure of acceptance and mindfulness for youth.
Dot-Probe Attention Task | 0, 3, and 6 mos
  Motivated attention task administered via computer to capture attentional bias toward emotional cues.

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Osher Center for Integrative Medicine, San Francisco, California, United States